CLINICAL TRIAL: NCT06796166
Title: The Impact of Artificial Intelligence-Supported Preoperative Education on Fear and Anxiety Levels in Total Mastectomy Patients: A Randomized Controlled Trial
Brief Title: The Impact of AI- Supported Education in Mastectomy Patient
Acronym: AI-ME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-13/548
Record Dates: First submitted 2024-12-09; First posted 2025-01-28 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Anxiety; Mastectomy; Patient Education as Topic; Artificial Intelligence (AI)
Keywords: artificial intelligence; fear of surgery; preoperative education; total mastectomy; breast cancer; surgical anxiety; patient education
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial with a parallel assignment design. Participants are randomly divided into two groups: an intervention group that receives AI-supported preoperative education and a control group that receives standard preoperative education. Both groups are assessed using validated tools to measure surgical fear and anxiety levels before and after the intervention. This design ensures that the impact of the AI-supported education is evaluated in comparison to the standard care.
Masking Description: This study is conducted as an open-label trial. Both participants and investigators are aware of the intervention assignments. The intervention group receives AI-supported preoperative education, while the control group receives standard preoperative education. Masking is not implemented as the nature of the intervention does not allow for blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Education Group (Experimental): Participants in this group will receive AI-supported preoperative education. This intervention involves an interactive, personalized digital education platform designed to reduce surgical fear and anxiety. The program includes detailed information about the surgical process, postoperative care, and emotional coping strategies. The AI platform allows patients to interactively ask questions and receive tailored responses.
  Interventions: Behavioral: AI-Supported Preoperative Education
- Traditional Education Group (Active Comparator): Participants in this group will receive standard preoperative education provided by healthcare professionals. The education consists of general information about the surgical process, postoperative care, and strategies for managing fear and anxiety. This group serves as a comparison to the experimental group receiving AI-supported education.
  Interventions: Behavioral: Standard Preoperative Education

INTERVENTIONS:
Behavioral: AI-Supported Preoperative Education — This intervention involves the use of a pre-trained AI-powered education platform designed to provide preoperative information to patients undergoing mastectomy. The program delivers structured, interactive education that includes details about the surgical process, postoperative care, and emotional coping strategies. The pre-trained AI system offers standardized responses to patient questions, ensuring consistency and clarity in the information provided, with the goal of reducing fear and anxiety.
  Arms: Digital Education Group
Behavioral: Standard Preoperative Education — This intervention consists of standard preoperative education provided by healthcare professionals. Patients receive general information about the surgical procedure, postoperative care, and strategies to manage fear and anxiety. The education is delivered in a traditional, face-to-face format without the use of AI or digital tools.
  Arms: Traditional Education Group

SUMMARY:
This study aims to evaluate the impact of artificial intelligence (AI)-supported preoperative education on fear and anxiety levels in patients undergoing total mastectomy. It is a randomized controlled trial involving two groups: one receiving AI-supported education and the other receiving standard preoperative education. The primary outcomes are to assess changes in surgical fear and anxiety levels. The study targets adult female patients diagnosed with breast cancer who are scheduled for total mastectomy.

DETAILED DESCRIPTION:
This study will aim to evaluate the impact of an artificial intelligence (AI)-supported preoperative education program on surgical fear and anxiety levels in patients undergoing total mastectomy. The study will be conducted using an experimental and randomized controlled design, with the control group receiving standard education and the experimental group receiving AI-supported education. The research will be carried out between 2024 and 2025 at the surgical unit of Acıbadem International Hospital.

Breast cancer continues to be the most common cancer type among women worldwide and a significant cause of morbidity and mortality. In Turkey, breast cancer is the most frequently diagnosed cancer among women and remains a leading cause of cancer-related deaths. Patients diagnosed with breast cancer often experience high levels of fear and anxiety, particularly during the surgical process. Literature suggests that between one-quarter and one-third of breast cancer patients develop anxiety during their treatment journey, with some cases progressing to depression.

Surgical fear and anxiety are critical factors that negatively impact the physical and psychological well-being of patients. Anxiety is often triggered by fear of death, uncertainties regarding the recovery process, and a perceived loss of control, while surgical fear focuses on potential physical harm or health risks associated with the surgery. Therefore, interventions to reduce fear and anxiety during the preoperative period will remain crucial.

Preoperative education is an effective method known to increase patient satisfaction and contribute positively to recovery. Traditional educational methods, such as written brochures and verbal instructions, are commonly used. However, these methods may not always be sufficient, particularly for patients experiencing high anxiety levels, as they may struggle to comprehend the information provided. At this point, the integration of technological innovations to make educational materials more interactive and effective has become a necessity. Artificial intelligence (AI) will stand out as one such innovative tool and is expected to enable healthcare professionals to deliver more effective patient education.

AI-supported educational programs will facilitate easier access to information for patients and provide a personalized learning experience. By complementing written and verbal materials, AI will offer interactive communication, allowing patients to ask questions and receive fast, clear, and satisfying responses. Additionally, such an approach will help reduce the workload of healthcare professionals, enabling them to reach a larger number of patients. Given that the number of nurses per capita in Turkey is significantly below the OECD average, these technological solutions will become even more important.

The primary objective of this study will be to evaluate the effect of an AI-supported preoperative education program on surgical fear and anxiety in total mastectomy patients. The research will adopt a randomized controlled design. Standard education will be provided to the control group, while interactive AI-supported education will be offered to the experimental group via a tablet. The educational content will cover topics such as the operating room environment, invasive procedures, deep breathing and respiratory exercises, spirometer use, postoperative recovery areas, surgical drains, wound care, mobilization, and professional nursing care.

A total of 40 patients will be included in the study, and participants will be randomized equally into experimental (AI-supported education) and control (standard education) groups. Data collection tools will include a Demographic Information Form, the State-Trait Anxiety Inventory (STAI), and the Surgical Fear Questionnaire (SFQ). Data will be analyzed using the SPSS program, with statistical tests such as independent t-tests, chi-square tests, and ANOVA applied to evaluate the differences between groups.

The expected results will show that AI-supported education is an effective method for reducing surgical fear and anxiety. This method is anticipated to save time for healthcare professionals while providing personalized, fast, and continuous education, ultimately improving patient satisfaction. The strengths of the study will include being among the first to test AI-supported education in mastectomy patients and determining the sample size through power analysis. However, limitations may include a small sample size and the study being conducted at a single hospital, which may restrict generalizability.

The research will be conducted with the necessary approvals from ethics committees and hospital administration. Participants' privacy will be safeguarded, and voluntary participation will be ensured. It is expected that AI-supported educational programs will prove to be an effective tool for both healthcare professionals and patients. These findings will serve as an important guide for restructuring educational and support practices for patients in the preoperative period.

ELIGIBILITY:
Inclusion criteria:

* Literate female patients
* Patients who will undergo total mastectomy surgery
* Patients diagnosed with breast cancer
* Patients who are over 18 years of age
* Patients who agree to participate in the study and from whom written consent has been obtained will be included in the study.

Exclusion criteria:

* Patients who cannot understand or communicate in Turkish
* Patients with active psychiatric disorders (e.g., major depression, bipolar disorder, schizophrenia)
* Patients with advanced hearing or vision problems
* Patients with mental disabilities
* Patients who have previously participated in a similar training program will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is limited to female participants because it focuses on conditions and interventions specific to women, particularly those undergoing mastectomy for breast cancer treatment.
Enrollment: 40 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Surgical Fear Questionnaire / SFQ | The scales will be administered twice: 15 minutes before the preoperative education session and 15 minutes after the preoperative education session.
  This outcome evaluates the change in surgical fear levels among participants using the Surgical Fear Questionnaire (SFQ).The scale consists of 8 items rated on an 11-point Likert scale ranging from 0 ("Not afraid at all") to 10 ("Very afraid"). It has two subdimensions, each consisting of 4 items, assessing the source of fear: Items 1-4 evaluate fear related to the short-term outcomes of surgery, while Items 5-8 evaluate fear related to the long-term outcomes. Subscale scores are calculated by summing the scores of the 4 items in each dimension, and the total scale score is obtained by summing the two subscale scores. Subscale scores range from 0 to 40, and the total scale score ranges from 0 to 80. Higher scores indicate higher levels of surgical fear.
State-Trait Anxiety Inventory /STAI | The scales will be administered twice: 15 minutes before the preoperative education session and 15 minutes after the preoperative education session.
  The State-Trait Anxiety Inventory (STAI) is a 20-item scale designed to measure temporary (state) and persistent (trait) anxiety levels. Anxiety is described as an emotional response to actual danger or threats in the environment or as a personality trait with individual differences. The STAI was developed as a self-assessment tool to evaluate the type and level of anxiety.
  The scale uses a 4-point Likert system, ranging from "Not at all" to "Completely." Twenty items assess state anxiety, while the other 20 items assess trait anxiety. Scores range from 20 to 80, with higher scores indicating higher anxiety levels. A score of 0-19 indicates no anxiety, 20-39 indicates low anxiety, 40-59 indicates moderate anxiety, and 60-80 indicates high anxiety. The Trait Anxiety Scale measures the tendency for persistent anxiety in daily life.

SECONDARY OUTCOMES:
Introductory Information Form | Before the Education
  In the study, the Introductory Information Form, consisting of 17 questions, is a data collection tool developed by the researcher. It includes information about the patients' socio-demographic characteristics (age, gender, marital status, education level, employment status, income level, occupation, and social security) and health history (current diagnosis and date, previous surgical experiences, and the presence of other health problems).

CONTACTS AND LOCATIONS:
Overall Officials: Mahmut DAGCI, PhD, Principal Investigator — Bezmialem Foundation University
Locations (1):
- Acibadem International Hospital, Istanbul, Bakirköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the sensitive nature of the data and privacy considerations for patients undergoing total mastectomy. Additionally, the institutional policies do not require sharing of IPD for this type of study.

REFERENCES:
- [Background] Biswas S. ChatGPT and the Future of Medical Writing. Radiology. 2023 Apr;307(2):e223312. doi: 10.1148/radiol.223312. Epub 2023 Feb 2. No abstract available. PMID 36728748
- See also: Provides global cancer statistics and projections, focusing on breast cancer — https://gco.iarc.fr/tomorrow/en/dataviz/isotype?cancers=20